CLINICAL TRIAL: NCT01457300
Title: Outcome of Multi-Disciplinary, Structured Rehabilitation of Older People in an Inpatient District Rehabilitation Centre Versus Standard Primary Health Care Rehabilitation - An Open Comparative Observational Stdy
Brief Title: Outcome of Rehabilitation of Older People in Primary Health Care
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: Norwegian Medical Association (Other)
Responsible Party: Principal Investigator, Inger Johansen, MD, PhD-student, University of Oslo
Other Study IDs: PHC rehab older people
Record Dates: First submitted 2011-10-12; First posted 2011-10-21 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Stroke; Hip Fractures; Osteoarthritis; Chronic Disease
Keywords: Rehabilitation outcome; Aged; Aged, 80 and over; Activities of daily living
MeSH Terms: conditions — Stroke; Hip Fractures; Osteoarthritis; Chronic Disease | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- District Rehabilitation Centre (Model 1): Patients admitted to Primary Health Care Rehabilitation, either Post-Acute from the Same District General Hospital or Directly from their Homes. They were recruited continuously at Entrance to the Rehabilitation Centre.
  Interventions: Other: Rehabilitation
- Standard PHC Rehabilitation (Model 2): Patients admitted to Standard Primary Health Care (PHC) Rehabilitation, either Post-Acute from the Same District General Hospital or Directly from their Homes. They were recruited Continuously at Entrance to the Short Term Rehabilitation Beds in Nursing Homes or at the Beginning of Rehabilitation in their Own Homes.

INTERVENTIONS:
Other: Rehabilitation — Model 1: Regular Assessment of Rehabilitation Goal, Rehabilitation Plan, Weekly Multi-Disciplinary Evaluation and Adjustment of Plan, Regular use of Measurement Scales, Regular Dialog between Personnel, Patient and Relatives. Model 2: More Occasional use of the Listed Activities. Model 1 and Model 2: Physical Training and Functional ADL Training, in Groups, One by One or Self-Training.
  Groups: District Rehabilitation Centre (Model 1)

SUMMARY:
The Outcome of Multi-Disciplinary, Structured Rehabilitation of Older People in a District Inpatient Rehabilitation Centre is better than in a Standard Primary Health Care Rehabilitation Programme in Short Term Beds in Nursing Homes.

ELIGIBILITY:
Inclusion Criteria:

* Both Genders
* Age=>65 Years
* Diagnoses: Stroke, Hip Fractures, Osteoarthritis, Chronic, slowly progressing Diseases, Functional Decline due to Old Age, Functional Decline due to Long Hospital Stay
* Assessed to have a Rehabilitation Potential

Exclusion Criteria:

* Age<65 Years
* Patietns with Highly Progressive Diseases
* Sunnaas ADL Index<10
* MMSE<18
* Deeply Depressed Patients with no Initiative
* Patients with Speech Dyspnoea
* Patients with unstable Angina Pectoris
* Patients with not diagnosed Cardiac Arrythmias

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The Study Populations were Disabled Older People (=>65years), with a need for Rehabilitation either Post-Acute after Hospitalisation or admitted Directly from their Own Homes and living within the Geographically small County of Vestfold, Norway.
Sampling Method: Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2006-06; Primary Completion 2009-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in Sunnaas ADL Index | Change from Baseline in Sunnaas ADL Index at End of Rehabilitation. Change from End of Rehabilitation in Sunnaas ADL Index at 3 months. Change from End of Rehabilitation in Sunnaas ADL Index at 18 Months
  Sunnaas ADL Index measures 12 Activities of Daily Life. Each Activity has a Score from 0-3, where 0=totally dependent and 3=independent. The Total Max Score of 36 means Totally Independent.

SECONDARY OUTCOMES:
Change in Umea Life Satisfaction Checklist | Change from End of Rehabilitation in Umea Life Satisfaction Checklist at 3 Months after Rehabilitation.
  A Simple and Validated Questionnaire, testing Life Satisfaction. We chose Two of the Questions: LSCa: How satisfied are you with your Life in general? LSCb: How satisfied are you with your Ability to manage your Self-Care? The Scores are 1-3=not satisfied and 4-6=satisfied
Mini Mental Status Evaluation=MMSE | MMSE Recorded Two Weeks into Rehabilitation
  MMSE measures Cognitive Function. Scores are from 0-30, where 30 indicates no Cognitive Problems.
Symptom Check List 10=SCL10 | SCL10 recorded at two Weeks into Rehabilitation
  SCL10 is a Questionnaire mapping Emotional Health during the Previous Week, particularly Anxiety and Depression. SCL-10 comprises Ten Questions with Scores from 1-4. The Final Score is the Total Score sum divided by Ten. Scores>1.85 indicate Severe Emotional Problems
Home Care Services | Change from End of Rehabilitation in Home Care Services at Three Months after Rehabilitation
  The care scores were: 1:0 hour/week, 2:>0-3 hours/week, 3:>3-6 hours/week, 4:>6-9 hours/week, and 5:>9 hours/week.
Informal Care from Relatives | Change in Informal Care from relatives from End of Rehabilitation at Three Months after Rehabilitation
  Care Scores: 1:0 Hour/Week, 2:>0-3 Hours/Week, 3:>3-6 Hours/Week, 4:>6-9 Hours/Week, and 5:>9 Hours/Week.

CONTACTS AND LOCATIONS:
Overall Officials: Inger Johansen, MD, Principal Investigator — University of Oslo; Mette Brekke, MD, PhD, Study Chair — University of Oslo
Locations (2):
- Norway (2):
  - Department of General Practice/General Practice Research Unit, Institute of Health and Society, University of Oslo, Oslo, Oslo County
  - Prestelokka Rehabilitation Centre, Stavern, Vestfold

REFERENCES:
- [Result] Johansen I, Lindbaek M, Stanghelle JK, Brekke M. Effective rehabilitation of older people in a district rehabilitation centre. J Rehabil Med. 2011 Apr;43(5):461-4. doi: 10.2340/16501977-0792. PMID 21390482
- [Derived] Johansen I, Lindbak M, Stanghelle JK, Brekke M. Independence, institutionalization, death and treatment costs 18 months after rehabilitation of older people in two different primary health care settings. BMC Health Serv Res. 2012 Nov 14;12:400. doi: 10.1186/1472-6963-12-400. PMID 23150906